CLINICAL TRIAL: NCT02258828
Title: An Open-Label Trial of Memantine for Cognitive Impairment in Patients With Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sriram Ramaswamy (U.S. Federal Agency)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Sriram Ramaswamy, STAFF PSYCHIATRIST, VA Nebraska Western Iowa Health Care System
Organization: VA Nebraska Western Iowa Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00255
Record Dates: First submitted 2014-10-02; First posted 2014-10-08 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental): Subjects initially received memantine 5 mg once daily, which was increased weekly by 5 mg/day in divided doses to a dose of 20 mg/day
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Patient received matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Subjects initially received memantine 5 mg once daily, which was increased weekly by 5 mg/day in divided doses to a dose of 20 mg/day
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
Twenty six veterans with PTSD and cognitive impairment received 16 weeks of memantine in an open label fashion. Cognition was assessed using the Spatial Span, Logical Memory I, and Letter-Number Sequencing subtests of the Wechsler Memory Scale III (Third edition) and the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). RBANS measures attention, language, visuospatial skills, and immediate and delayed memories. The Clinician Administered PTSD Scale (CAPS), Hamilton Depression Scale (HAM-D), Hamilton Anxiety Scale (HAM-A), Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q), and Sheehan Disability Scale (SDS) were used to assess improvement in PTSD symptoms, as secondary outcome measures.

DETAILED DESCRIPTION:
Participants were recruited from the Omaha Veterans Affairs Medical Center following local IRB approval. We obtained written consent from all the subjects who were recruited in the study. Veterans between the ages of 19 and 65 years with chronic PTSD (diagnosis for >6 months) attributable to military combat exposure were included in the study. Patients were required to be clinically stable on their psychotropic medication regimen for at least three months prior to study entry. In addition to meeting DSM-IV criteria for PTSD and endorsing subjective complaints of memory difficulties, patients had to score least one standard deviation below the mean performance of a standardized, age- and sex-matched population on the Spatial Span, Logical Memory I, and Letter-Number Sequencing subtests of the Wechsler Memory Scale III (Third edition) for study entry. Patients with a history of dementia, schizophrenia, bipolar disorder, traumatic brain injury, and seizure were excluded. Patients with any history of alcohol or illicit drug abuse or dependence within the past one month were excluded. Patients requiring concomitant treatment with drugs with potential effects on the glutamergic system, such as amantadine,dextromethorphan, or carbonic anhydrase inhibitors, were excluded.

Subjects initially received memantine 5 mg once daily, which was increased weekly by 5 mg/day in divided doses to a dose of 20 mg/day. Memory was assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) [Randolph, 1998] using both forms A and B at baseline, end of week 8, and end of week 16. The RBANS is composed of 10 subtests that yield a total score and five index scores: immediate memory, visuospatial/constructional, language, attention, and delayed memory. Each index score has a normal mean of 100 and standard deviation of 15 based on the performance of a standardization sample matched to the U.S. Census on sex, ethnicity, and level of education. Alternative forms of the RBANS (Forms A and B) were used to avoid bias due to practice effects. We administered Clinician Administered PTSD Scale (CAPS), Hamilton Depression Scale (HAM-D), Hamilton Anxiety Scale (HAM-A), Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q), and Sheehan Disability Scale (SDS) to assess the secondary measures. Changes in the scores over time with repeated measures were estimated with mixed-effects models. The primary outcome measures of interest were index and percentile scores in RBANS total and subscale scores. The repeated measures model included visit (as a categorical variable) as a fixed effect. An unstructured covariance matrix was used to fit the within patient repeated measures effect. Tukey's method was used to compare pair-wise means.

Secondary outcome measures, CAPS, HAM-A, HAM-D, Q-LES-Q, and SDS, were analyzed similarly to the RBANS with repeated measures models. P-values less than 0.05 are considered to be statistically significant. SAS software version 9.1 (SAS Institute, Cary, NC) was used for the analysis

ELIGIBILITY:
Inclusion Criteria:

1. Patients, men and women between 18 and 65 years of age, inclusive.
2. Patients with diagnosis of Posttraumatic Stress Disorder (309.81) for at least 6 months, as determined by the Structured Clinical Interview for DSM-IV Axis 1 Disorders (SCID).
3. Patients with a score of at least 1 standard deviation below the mean on the Spatial Span, Logical Memory I and Letter-Number Sequencing subtest's of the Wechsler Memory Scale III (Third edition).
4. Patients, who are able to comprehend and satisfactorily comply with protocol requirements and have an ability to read and write English,
5. Patients, who signed the written informed consent given prior to entering any study procedure.
6. Patients must be clinically stable on their medications for past three months

Exclusion Criteria:

1. Patients with a concurrent DSM-IV Axis I or Axis II diagnosis in any of the following categories:

   * 1.1. Delirium, Dementia, Amnestic and other Cognitive disorders
   * 1.2. Mental Retardation
   * 1.3. Lifetime Schizophrenia and other Psychotic Disorders
   * 1.4. Lifetime Bipolar I Disorder
   * 1.5. Alcohol or Substance Dependence or Abuse (excluding nicotine) in one month prior to the Screening Visit
   * 1.6. Any other concurrent Axis I Disorder (including Major Depressive Disorder) must be secondary to the primary diagnosis of PTSD.
2. Patients with a score of less than 1 standard deviation below the mean on the Spatial Span, Logical Memory I and Letter-Number Sequencing subtest's of the Wechsler Memory Scale III at the screening visit.
3. Patients with a history of treatment with cholinesterase inhibitor drugs like donezepil, galantamine or rivigstamine.
4. Patients with a history of intolerance or hypersensitivity to memantine.
5. Patients with a history of seizures and traumatic head injury.
6. Patients requiring concomitant treatment amantadine or dextromethorphan or carbonic anhydrase inhibitors.
7. Patients who based on history or mental status examination have a significant risk of committing suicide.
8. Patients who are homicidal or violent and who are in the Investigator's opinion in significant imminent risk of hurting others.
9. Patients with a positive urine drug screen, for drugs of abuse.
10. Patients who have participated in any clinical trial within one month prior to the Screening Visit, or in a clinical trial involving a psychotropic medication within the 3 months prior to the Screening Visit.
11. Patients who have a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial.
12. Patients with any current malignancy, or any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease (including any form of epilepsy). If there is a history of such disease but the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
13. Patients whose laboratory values at the Screening visit will be 2 times greater than ULN.
14. Patients who require concomitant therapy with any prohibited prescription or over-the-counter medication.
15. Patients who are unable to speak, read, and understand English or are judged by the investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits.
16. Women patients who are pregnant, planning to become pregnant, or if of childbearing potential, not using an acceptable method of birth control.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
RBANS | 16 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Ramaswamy, MD, Principal Investigator — Department of Veterans Affairs/NWIHCS
Locations (1):
- Omaha Veterans Affairs Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes